CLINICAL TRIAL: NCT02393690
Title: Randomized Double-Blind Phase II Study of Radioactive Iodine (RAI) in Combination With Placebo or Selumetinib for the Treatment of RAI-Avid Recurrent/Metastatic Thyroid Cancers
Brief Title: Iodine I-131 With or Without Selumetinib in Treating Patients With Recurrent or Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RU241306I; NCI-2015-00277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-008494; RU241306I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-03-19 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Thyroid Gland Carcinoma; Poorly Differentiated Thyroid Gland Carcinoma; Recurrent Thyroid Gland Carcinoma; Stage IV Thyroid Gland Follicular Carcinoma AJCC v7; Stage IV Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVA Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVA Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVB Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVB Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVC Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVC Thyroid Gland Papillary Carcinoma AJCC v7
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Iodine-131; AZD 6244

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (selumetinib, iodine I-131) (Experimental): Patients receive selumetinib PO BID starting on week 1, day 1 and continuing through 2 days after iodine I 131 therapy has been administered. Approximately 3 weeks after beginning treatment with selumetinib, patients receive iodine I-131 PO.
  Interventions: Radiation: Iodine I-131; Drug: Selumetinib
- Arm II (placebo, iodine I-131) (Active Comparator): Patients receive placebo PO BID starting on week 1, day 1 and continuing through 2 days after iodine I-131 therapy has been administered. Approximately 3 weeks after beginning treatment with placebo, patients receive iodine I-131 PO.
  Interventions: Radiation: Iodine I-131; Other: Placebo Administration

INTERVENTIONS:
Radiation: Iodine I-131 — Given PO
  Other Names: 131-Iodine; Bound Iodide I-131; I 131; I-131; Iodide I-131; Iodide, I-131; Iodine 131; Iodotope; Iodotrope
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo, iodine I-131)
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244
  Arms: Arm I (selumetinib, iodine I-131)

SUMMARY:
This phase II trial studies how well iodine I-131 works with or without selumetinib in treating patients with thyroid cancer that has returned (recurrent) or has spread from where it started to other places in the body (metastatic). Many thyroid cancers absorb iodine. Due to this, doctors often give radioactive iodine (iodine I-131) alone to treat thyroid cancer as part of standard practice. It is thought that the more thyroid tumors are able to absorb radioactive iodine, the more likely it is that the radioactive iodine will cause those tumors to shrink. Selumetinib may help radioactive iodine work better in patients whose tumors still absorb radioactive iodine. It is not yet known whether iodine I-131 is more effective with or without selumetinib in treating thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the response rate at 6 months following treatment with 131I (iodine I-131) in combination with placebo or selumetinib for radioactive iodine-avid (RAIA) recurrent and/or metastatic thyroid cancer.

SECONDARY OBJECTIVES:

I. To determine the best overall response following treatment with 131I in combination with placebo or selumetinib for RAIA recurrent and/or metastatic thyroid cancer.

II. To compare the progression-free survival of patients with RAIA recurrent and/or metastatic thyroid cancer treated with 131I in combination with placebo or selumetinib.

III. To compare serum thyroglobulin changes for patients with RAIA recurrent and/or metastatic thyroid cancer treated with 131I in combination with placebo or selumetinib.

IV. To evaluate the safety and tolerability of 131I in combination with placebo or selumetinib for patients with RAI-avid recurrent and/or metastatic thyroid cancer.

CORRELATIVE OBJECTIVE:

I. To explore the genomic and transcriptomic landscape of RAIA tumors for signatures that correlate to therapeutic benefit achieved with 131I in combination with placebo or selumetinib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive selumetinib orally (PO) twice daily (BID) starting on week 1, day 1 and continuing through 2 days after iodine I-131 therapy has been administered. Approximately 3 weeks after beginning treatment with selumetinib, patients receive iodine I-131 PO.

ARM II: Patients receive placebo PO BID starting on week 1, day 1 and continuing through 2 days after iodine I-131 therapy has been administered. Approximately 3 weeks after beginning treatment with placebo, patients receive iodine I-131 PO.

After completion of study treatment, patients are followed up at 1 and 3 months, every 3 months for 12 months, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent and/or metastatic thyroid cancer
* Histological or cytological confirmation of thyroid carcinoma of follicular origin (including papillary, follicular, or poorly differentiated subtypes and their respective variants); NOTE: medullary and anaplastic thyroid cancers are excluded; Hurthle cell carcinomas are excluded (defined as having an invasive tumor composed of > 75% oncocytic [Hurthle] cells lacking the nuclear features of papillary carcinoma, tumor necrosis, and marked mitotic activity); patients with oncocytic (Hurthle cell) variants of papillary thyroid carcinoma (defined as a tumor composed of a majority of oncocytic [Hurthle] cells having the nuclear features of papillary carcinoma) are eligible to participate
* RAI-avid lesion on a radioiodine scan (a diagnostic, post-therapy, or post-ablation scans) performed =< 24 months prior to registration, which suggests that therapy with 131I is justifiable in the judgment of the investigator
* Clinically or radiographically evident structural disease; patients with measurable disease and those with only non-measurable ("non-target") structural disease (according to modified Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1 criteria) are eligible;

NOTE 1: Modification of the RECIST v1.1 measurable disease criteria includes a change in the definition of what is considered a measurable malignant lymph node; a malignant lymph node is considered measurable if any of the following apply:

* It is noted to be RAI-avid on radioactive iodine imaging (diagnostic or post-therapy whole body scans acceptable) and it measures >= 1 cm in the long axis,
* It is pathologically proven to be involved with thyroid cancer (by cytology or pathology) and it measures >= 1 cm in the long axis, or
* Its short axis is >= 1.5 cm when assessed by computed tomography (CT) scan NOTE 2: Patients only with biochemical evidence of disease without structural evidence of cancer are not eligible for this study

  * For patients with non-measurable, structural disease the following must apply:
* Undetectable thyroglobulin antibody AND
* A serum thyroglobulin of 10 ng/ml or greater in the context of suppressed thyroid-stimulating hormone (TSH) (TSH =< 0.4 mcU/ml) =< 28 days prior to study registration; use of any thyroglobulin assay is allowed, though all serum thyroglobulin measurements for study purposes must be conducted with the same thyroglobulin assay

  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
  * Able to swallow and retain orally-administered medication with no clinically significant gastrointestinal abnormalities that may alter absorption
  * Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to randomization)
  * Platelet count >= 100,000/mm^3 (obtained =< 28 days prior to randomization)
  * Hemoglobin > 9.0 g/dL (obtained =< 28 days prior to randomization)
  * Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 28 days prior to randomization)
  * Aspartate transaminase (AST) =< 2.5 x ULN (or =< 5 x ULN in presence of liver metastases) (obtained =< 28 days prior to randomization)
  * Creatinine =< 1.5 mg/dL OR calculated creatinine clearance of >= 50 ml/min by either the Cockcroft-Gault formula or 24-hours urine collection analysis (obtained =< 28 days prior to randomization)
  * Negative pregnancy test performed =< 7 days prior to registration for women of childbearing potential only
  * Provide informed written consent
  * Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Note: during the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up

  * Willing to provide mandatory archival tumor tissue (block or minimum of 30 unstained slides from a primary or recurrent/metastatic thyroid cancer) for correlative research purposes; NOTE: patients with less archival tumor tissue available may still be eligible for the study after discussion with Academic and Community Cancer Research United (ACCRU); receipt of archival tumor tissue is not required for study registration and initiation of therapy
  * Willing to provide mandatory blood samples for correlative research purposes

Exclusion Criteria:

* 131I therapy =< 6 months prior to registration; Note: 131I administered solely for diagnostic purposes is not considered 131I therapy
* External beam radiation therapy =< 28 days prior to registration; note: previous treatment with radiation is allowed if the investigator judges it will not compromise patient safety on the study
* Having been treated with a total cumulative (lifetime) 131I therapeutic activity > 800 mCi (excluding 131I activity administered for diagnostic scans)
* Treatment with chemotherapy or targeted therapy (e.g. tyrosine kinase inhibitor) =< 28 days prior to registration
* Prior exposure to mitogen-activated protein kinase kinase (MEK), RAS, or RAF inhibitors (note: previous exposure to sorafenib is allowed) OR history of hypersensitivity to selumetinib, thyrotropin alpha (Thyrogen), or any excipient agents
* Unresolved toxicity > Common Terminology Criteria for Adverse Events (CTCAE) grade 2 from previous anti-cancer therapy, except for alopecia
* Cardiac conditions as follows:

  * Uncontrolled hypertension (blood pressure [BP] >=150/95 mmHg despite medical therapy)
  * Left ventricular ejection fraction < 55% measured by echocardiography
  * Atrial fibrillation with a ventricular rate > 100 beats per minute (bpm) on electrocardiogram (ECG) at rest
  * Symptomatic heart failure (New York Heart Association [NYHA] grade II-IV)
  * Prior or current cardiomyopathy
  * Severe valvular heart disease
  * Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy)
  * Acute coronary syndrome =< 6 months prior to registration
* Ophthalmological conditions as follows:

  * Intra-ocular pressure > 21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure)
  * Current or past history of central serous retinopathy or retinal vein occlusion
* Symptomatic or untreated leptomeningeal disease, brain metastasis, or spinal cord compression
* Unable to follow a low iodine diet or requiring medication with high content in iodide (e.g., amiodarone)
* Received iodinated intravenous contrast within =< 2 months of registration; avoidance of iodinated oral contrast is also preferred but not strictly required for study enrollment; NOTE: those who have had iodinated intravenous contrast within this time frame may still be eligible if a urinary iodine analysis reveals that excess iodine has been cleared (defined as urinary iodine documented to be < 300 mcg/day by either a spot urinary iodine or 24-hour urinary iodine measurement)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hepatitis B infection, hepatitis C infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm. (NOTE: Performance of investigational 124I PET/CT scans is allowed prior to and during conduct of this study)
* Other active malignancy =< 2 years prior to registration that will interfere with conduct of this trial; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, patients must not be receiving other specific treatment (chemotherapy, hormonal therapy, radiation) for their cancer
* Not willing to discontinue use of supplemental vitamin E

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Ho, Principal Investigator — Academic and Community Cancer Research United
Locations (11):
- United States (11):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Hoag Memorial Hospital, Newport Beach, California
  - University of Colorado Hospital, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Selumetinib, Iodine I-131): Patients receive 75 mg selumetinib PO BID starting on week 1, day 1 and continuing through 2 days after iodine I 131 therapy has been administered. Approximately 3 weeks after beginning treatment with selumetinib, patients receive iodine I-131 PO.
Period: Overall Study
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
Started | 28 | 30
Completed | 28 | 29
Not Completed | 0 | 1
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients registered to protocol treatment are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Median (Full Range); unit: years] | 62 [20 to 78] | 61 [24 to 83] | 62 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 19 | 23 | 42
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Response at 6 Months
Description: A patient will be classified as a responder if they have a partial or complete response at the 6-month time point when compared to the baseline, pre-study radiologic scan(s). A Complete Response (CR) is defined as the disappearance of all target lesions and thyroglobulin measured to be less than 0.2 ng/ml. A Partial Response (PR) is defined as at least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the long or short axis of all the target lymph nodes (depending on which axis is being used for assessments) at current evaluation) taking as reference the baseline sum of dimensions (BSD).
  >
  > A patient will be classified as a responder if they have a partial or complete response at the 6-month time point. The proportion of patients with a response will be calculated and compared between the 2 Arms using a Fisher's Exact test.
Time Frame: At 6 months
Population: All patients that began protocol treatment and were evaluable for this endpoint are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
Number analyzed (Participants) | 28 | 29
Participants | 7 | 2
Statistical Analysis 1: Comparison: Arm I (Selumetinib, Iodine I-131) vs Arm II (Placebo, Iodine I-131); Test type: Superiority; p = 0.0787, Fisher Exact

2. Secondary Outcome: Overall Response Rate
Description: The best overall response rate will be compared between the two arms. This comparison will be done using a Fisher exact test. For a patient to be classified as a response, they need a partial or complete response that is confirmed at least 4 weeks later anytime during the study.
Time Frame: 2 years
Population: All patients that began protocol treatment and were evaluable for this endpoint are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
Number analyzed (Participants) | 28 | 29
Participants | 7 | 2
Statistical Analysis 1: Comparison: Arm I (Selumetinib, Iodine I-131) vs Arm II (Placebo, Iodine I-131); Test type: Superiority; p = 0.0787, Fisher Exact

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Time Frame: 2 years
Population: All patients that began protocol treatment and were evaluable for this endpoint are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
Number analyzed (Participants) | 28 | 29
months | 19 [12.4 to NA] — The upper limit of the confidence interval is not able to be estimated due to a low number of events. | 10.2 [6.8 to NA] — The upper limit of the confidence interval is not able to be estimated due to a low number of events.
Statistical Analysis 1: Comparison: Arm I (Selumetinib, Iodine I-131) vs Arm II (Placebo, Iodine I-131); Test type: Superiority; p = 0.1764, Log Rank

4. Secondary Outcome: Changes in Serum Thyroglobulin Levels
Description: Changes in serum thyroglobulin levels will be compared between the 2 treatment arms by 6 month response using the Wilcoxon Rank-Sum test.
Time Frame: 6 months
Population: All patients that began protocol treatment and were evaluable for this endpoint are included.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
Number analyzed (Participants) | 28 | 29
percent change from baseline | -29.1 (50.36) | 4.3 (61.28)
Statistical Analysis 1: Comparison: Arm I (Selumetinib, Iodine I-131) vs Arm II (Placebo, Iodine I-131); Test type: Superiority; p = 0.0756, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Incidence of Adverse Events
Description: The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The number and percentage of patients experiencing grade 3+ adverse events will be compared between the 2 treatment arms.
Time Frame: 2 years
Population: All patients that began protocol treatment and were evaluable for this endpoint are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
Number analyzed (Participants) | 28 | 29
Participants | 6 | 1

6. Other Pre Specified Outcome: Genomic and Transcriptomic Landscape of Radioactive Iodine-avid (RAIA) Tumors
Description: Will explore the genomic and transcriptomic landscape of RAIA tumors for signatures that correlate to therapeutic benefit achieved in patients with RAI-avid recurrent and/or metastatic thyroid cancer treated with 131I in combination with placebo or selumetinib. Exploratory analysis will include correlating response to tumor genotypes. Descriptive statistics and graphical techniques will be used to summarize this data by treatment arm.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each 28 day cycle. The max number of cycles taken was 8.
Description: Adverse events were collected at the end of each 28 day cycle. The max number of cycles taken was 8.
Arm/Group | Arm I (Selumetinib, Iodine I-131) | Arm II (Placebo, Iodine I-131)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/30
Other Adverse Events (participants affected / at risk) | 28/28 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Selumetinib, Iodine I-131) (N=28) | Arm II (Placebo, Iodine I-131) (N=30)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Selumetinib, Iodine I-131) (N=28) | Arm II (Placebo, Iodine I-131) (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 7 (11) | 3 (5)
Retinopathy (Eye disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (19) | 10 (16)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (16) | 9 (12)
Vomiting (Gastrointestinal disorders) | 4 (5) | 0 (0)
Fatigue (General disorders) | 20 (50) | 19 (41)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 12 (22) | 3 (5)
Alanine aminotransferase increased (Investigations) | 7 (12) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (16) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (15) | 1 (1)
Platelet count decreased (Investigations) | 9 (20) | 5 (10)
Weight loss (Investigations) | 1 (1) | 3 (5)
White blood cell decreased (Investigations) | 9 (26) | 4 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (15) | 5 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 14 (24) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (21) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 16 (44) | 15 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT02393690/Prot_SAP_ICF_000.pdf